CLINICAL TRIAL: NCT03616015
Title: Intestinal Dysbiosis and Immune Reconstitution After Allogeneic Hematopoietic Cell Transplantation
Brief Title: Dysbiosis and Immune Reconstitution After Allo-HSCT
Acronym: PARI-DYS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-A00676-49
Record Dates: First submitted 2018-07-19; First posted 2018-08-06 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: HSCT; intestinal dysbiosis; immune reconstitution
MeSH Terms: interventions — Blood Specimen Collection; Test Anxiety Scale; Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient (Experimental): For all patients included in the study, the following interventions will be performed :
  * several blood samples (quantity collected requiring classification of this study as interventional according to French law)
  * several fecal samples
  * anxiety tests
  * stress tests
  Interventions: Biological: blood samples; Biological: fecal samples; Behavioral: Anxiety test; Behavioral: Stress test

INTERVENTIONS:
Biological: blood samples — 20 to 30 ml of blood sample (D0, D15, D30, D60, D90, D180, Y1, Y2)
Biological: fecal samples — 1 g of feces (D-8, D0, D15, D30, D90)
Behavioral: Anxiety test — Test of Spielberger
Behavioral: Stress test — Test of Cohen

SUMMARY:
Preliminary (proof of concept), monocentric, interventional, prospective, non-randomized and analytic trial designed to simultaneously explore intestinal microbiota changes and early post-transplant immune reconstitution, and to correlate biological data with clinical data (antibiotics use, stress level, GVHD).

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is the major curative therapeutic approach for hematologic neoplasms. After HSCT, patients have a compromised GI mucosal barrier and an altered microbiota, also called dysbiosis. The later could be due to conditioning or use of broad-spectrum antibiotics, and could be accentuate by stress encountered by patients during their therapy management. Recent data have shown that alterations in the intestinal flora are associated with bad outcome, particularly with graft-versus-host disease (GVHD), bacteremia, and reduced overall survival post-transplantation. How intestinal bacteria can modulate the risk of relapse after HSCT is yet unknown. The scientists hypothesize that the variation of some bacterial taxa may influence post-transplant immune reconstitution, particularly invariant Natural Killer T cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years affiliated to a social security system
* Patients followed at the hospital of Nancy for a allogeneic hematopoietic cell transplantation (HLA matched donor)
* Graft of peripheral blood stem cell
* GVHD prophylaxis by ciclosporin and antilymphocyte serum +/- mycophenolate mofetil or methotrexate.

Exclusion Criteria:

* HIV+ patients
* Patients with active HBV or HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-12-04 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
quality of iNKT reconstitution after HSCT (good/poor) | Day 90,

SECONDARY OUTCOMES:
gut microbiota composition | Day 0, Day 15, Day 30, Day 90
  relative abundance of intestinal bacterial taxa
immune reconstitution after HSCT (other immune cells) | Day 15, Day 30, Day 60, Day 90, Day 180, Year 1, Year 2
  quantification of Tregs, MDSC, MAIT, T lymphocytes
GVH disease | Day 30, Day 60, Day 90
  yes/not
use of antibiotics | Day 0, Day 15, Day 30, Day 60, Day 90
  yes/not (molecules, delay, posology)
level of stress | Day -8, Day 15, Day 30, Day 90
  test of Cohen
level of anxiety | Day -8, Day 15, Day 30, Day 90
  test of Spielberger
quality of iNKT reconstitution after HSCT (good/poor) | Day 15, Day 30, Day 60, Day 180, Year 1, Year2

CONTACTS AND LOCATIONS:
Locations (1):
- RUBIO Marie-Thérèse, Vandœuvre-lès-Nancy, France